CLINICAL TRIAL: NCT02492633
Title: Prospective Evaluation of a Comprehensive Smoke-Free Public Housing Policy in a Multi-State Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Boston University (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, Vaughan Rees, Director of the Center for Global Tobacco Control; Lecturer on Social and Behavioral Sciences, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MAHHU0025-14
Record Dates: First submitted 2015-07-06; First posted 2015-07-08 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-08

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Smoke-free housing; Affordable housing; Second-hand smoke; Tobacco control
MeSH Terms: conditions — Smoking Cessation | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): The Standard Intervention will be offered to residents at all of Beacon Communities properties, regardless of the presence of this study.
  Interventions: Behavioral: Control
- Enhanced (Experimental): At a subset of 6 Beacon Communities properties, residents will receive an 'enhanced intervention' in addition to the 'standard intervention' that Beacon Communities is already providing.
  Interventions: Behavioral: Control; Behavioral: Intervention

INTERVENTIONS:
Behavioral: Control — The Standard Intervention will be offered to residents at all of Beacon Communities properties, regardless of the presence of this study. The standard intervention will be implemented as part of the smoke-free initiative roll out and will consist of: monthly articles in newsletters, re-usable shopping bag giveaways touting cessation messages, information provided via the property websites, and training of Residential Service Coordinators (RSCs) using the 8-session smoking cessation group training provided by the American Lung Association. The RSCs will offer group cessation counseling sessions for residents who would like support to quit smoking.
Behavioral: Intervention — At a subset of 6 Beacon Communities properties, residents will receive an 'enhanced intervention' in addition to the 'standard intervention' that Beacon Communities is already providing. The enhanced intervention will consist of the following:
  1. A web-based smoking cessation intervention via Facebook
  2. Enhanced gain-framed messaging communicated via several channels. Gain framed messages will incorporate themes of smoking cessation and policies which aim to distinguish from the vast 'library' of traditional messages which focus on loss-framing.
  3. A behavioral "nudge" designed to enhance public support for the smoke free policy, through personal adoption and adherence to the policy. This will be done by promoting a publicly viewable "pledge" program.
  Arms: Enhanced

SUMMARY:
The primary objective of this project is to evaluate the effectiveness of an enhanced intervention vs. a standard intervention to complement a comprehensive smoke-free policy, in a multi-site, privately managed affordable housing context.

DETAILED DESCRIPTION:
Beacon Communities, a private property management company, is unveiling a comprehensive smoking ban at all 52 of its properties. A multi-component, "enhanced" intervention designed to promote, strengthen, and maintain a smoke-free policy across public housing developments will be implemented prior to commencement of the smoke-free policy. The enhanced intervention will be tested against a standard intervention of educational materials and information on cessation options. This study will be open to residents at 12 Beacon Communities properties at which a Resident Service Coordinator (RSC) is located.

The primary objective of this project is to evaluate the effectiveness of enhanced intervention vs. standard intervention to support a comprehensive smoke-free policy, in a multi-site, privately managed affordable housing context. A further objective is to develop a toolkit of strategies for the large-scale implementation and maintenance of a smoke-free policy in multi-unit affordable housing developments. The toolkit will be the first to be developed directly from an extensive two-stage qualitative analysis and will apply the lessons learned in this study to provide a sustainable resource for property managers seeking to implement smoke-free policies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Able to speak English or Spanish
* A resident of Beacon Communities housing development (12 selected sites)
* Thinks that he/she will be living in his/her Beacon Community for at least the next 12 months

For Smokers:

* Have smoked cigarettes or e-cigarettes in the last week

For Non-Smokers:

* Self-reported exposure to secondhand smoke in the previous 2 months

Exclusion Criteria:

* Have another household member enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in cigarettes smoked in the home | 12 months
  Cigarettes smoked in the home (defined as self-reported number of cigarettes smoked in the home in past 30 days) at the 12-month follow up assessment, compared with pre-baseline level.

SECONDARY OUTCOMES:
Air quality | 12 months
  Indoor air quality will be measured using airborne nicotine concentration (ug/m3) at the 12-month follow up assessment, compared with pre-baseline level.
Change in motivation to quit smoking | 12 months
  Motivation to quit smoking (assessed by self-report on the 12-month follow up assessment), at 12 month follow-up, compared with pre-baseline level.

CONTACTS AND LOCATIONS:
Overall Officials: Vaughan Rees, PhD, Principal Investigator — Harvard TH Chan School of Public Health

IPD SHARING:
Plan to Share IPD: No